Official Title: Survivor Moms' Companion: A Perinatal Post-Traumatic Stress

Disorder Program

Unique Protocol ID: STUDY00007685

Date: 8/28/2023



## What is the Survivor Moms' Companion?

The Survivor Moms' Companion (SMC) is an education program for pregnant or postpartum women who have experienced abuse (either physically, sexually, or emotionally) when they are growing up. The SMC provides information about how past abuse and trauma can affect pregnancy and birth and provides you with a tutor to help you understand the material and support your learning.

# How can I sign up?

Participation in this program is completely voluntary. Whether or not you take part is completely up to you, and you can agree to take part and later change your mind. Your decision to participate will not be held against you. You will be assigned a SMC tutor at Buffalo Prenatal-Perinatal Network to help you through this program. Your SMC tutor will recommend you stop doing this program if you disclose a need for higher-priority services like domestic violence or mental health treatment, or if just isn't the right time for you to do this program. There is no cost to you for the program workbook materials or for the tutor sessions.

## What happens if I say yes, I want to be in this program?

The Survivor Moms' Companion consists of a series of 10 "modules" that are written specifically to address the needs of women who are survivors of abuse. You will be invited to read a minimum of 4 of the modules (one per week) and then discuss your reactions with a tutor who will be assigned to you in a weekly 30-minute phone call or in-person meeting. Additionally, we will ask you to do 2 surveys interviews, which each take about 30 minutes. The first survey takes place before you start reading the modules, and asks about traumatic symptoms you may have had. The second survey is similar to the first and takes place after you complete the modules and tutoring sessions. You will be paid a \$30 gift card for completing the first survey and \$40 gift card for completing the second survey. Some participants will begin this program right away, and some will begin in 6 weeks; you will be randomly assigned to begin right away or in 6 weeks' time. Your total participation in the program will be about between 6 and 10 weeks once you begin the program. All of the information you share with your tutor will be entered into a secure database that will not be connected in any way to your health care records and will not have any identifying information about you attached to it. Researcher Dr. Mickey Sperlich at the University at Buffalo School of Social Work will be analyzing this anonymous data as part of an ongoing effort to study the Survivor Moms' Companion program.

#### Is there any way being in this study could be bad for me?

There may be some risk or discomfort from your participation in this research. The risk comes from the sensitive topic of the interviews, which could cause distress or problems for you if we failed to keep this information confidential. Distress from the questions is rare. If you feel distress during the interview, the

IRB Approval Period HRPP Revision Date: September 17, 2015 research assistant who is asking the questions can help you with your feelings right then, and she can give you resources to contact for more help.

To protect the sensitive information you give us, we store all information about you securely: for instance, all documents with your identity on them are stored completely separately from the survey answers. Electronic documents are kept on a secure database that is password-protected. Only research team members can access these documents, and they will not have access to your identity in any way. The researchers who will be analyzing data have completed training on keeping research information confidential.

Another possible risk is that you may worry that you need to take part in order to be on good terms with the health care staff or mental health care staff at the clinic where you were recruited to the study. You can participate in the program and choose not to participate in the research. Your decision to participate or not will not affect any health care or mental health care you receive.

## Will being in this study help me in any way?

We hope that your participation will help you feel more confident as you move forward in your role as a new mother. But regardless of whether you experience such a benefit from being in this study, others may benefit because this research may show the program is helpful and it may become available for more women to use.

## What happens to the information collected for the research?

Dr. Sperlich plans to publish the results of this study about whether the SMC was effective in helping women survivors. We will not include any information that would identify you. Your privacy will be protected and your research records will be confidential. It is possible that other people may need to see the information you give us as part of the study, such as organizations responsible for making sure the research is done safely and properly like the University at Buffalo, government offices or the study sponsor. There are some exceptions to keeping confidentiality. If you tell us something that makes us believe that you or others may be physically harmed, we may report that information to the appropriate agencies.

#### What else do I need to know?

This research is being funded through prize money received from the National Institutes of Health. It has been reviewed and approved by an Institutional Review Board ("IRB"). If you have questions, concerns, or complaints, or think the research has hurt you, you may talk to them at (716) 888-4888 or email <a href="mailto:ub-irb@buffalo.edu">ub-irb@buffalo.edu</a>. You can also contact the SMC researcher Dr. Mickey Sperlich at (716) 645-9087, or email at <a href="mailto:msperlic@buffalo.edu">msperlic@buffalo.edu</a>. You may also contact the research participant advocate at 716-888-4845 or <a href="mailto:researchadvocate@buffalo.edu">researchadvocate@buffalo.edu</a>.

## How do I sign up?

To see if you are eligible for this study and to get started, please call our research office at: (716)-255-7691.